CLINICAL TRIAL: NCT04103723
Title: Impact of Premedication on Anxiety: a Multi-centre, Prospective Observational Cohort Study
Brief Title: Impact of Premedication on Anxiety
Acronym: Impact
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Ana Kowark, Consultant, RWTH Aachen University
Other Study IDs: 19-132
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Preoperative Anxiety
Keywords: Midazolam; Premedication; Preoperative anxiety; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with premedication: Patients receiving preoperative premedication with midazolam before surgery.
  Interventions: Procedure: Preoperative premedication
- patients without premedication: Patients without preoperative premedication before surgery.
  Interventions: Procedure: Preoperative premedication

INTERVENTIONS:
Procedure: Preoperative premedication — Every patient with or without a preoperative premedication with midazolam before surgery.

SUMMARY:
IMPACT aims to evaluate the clinical routine practice of premedication in German hospitals and to estimate the influence of premedication on anxiety reduction.

DETAILED DESCRIPTION:
Generalised premedication with benzodiazepines in all surgical patients has become questionable, regarding the risk-benefit assessment and the lack of evidence for this practice. One of the main justifications for premedication with benzodiazepines is its anxiolytic effect. Anxiety is associated with postoperative cognitive and behavioural changes, physiological reactions, increased need of anaesthetic drugs and altered perception of pain, mood swings, wound-healing problems and alteration of the immune system. However, several investigations revealed negative side-effects like dose-dependent sedation up to respiratory depression, prolonged extubation-time, impaired psychomotor function, paradox reactions, antegrade amnesia, increased pneumonia rates and postoperative delirium.

In Germany midazolam is the most frequently administered premedication. A survey revealed that about one third of the German hospitals withhold a premedication in patients older than 74 years.

The evidence for this practice, as well as the indiscriminate preoperative premedication for all adult patients is low.

The investigators aim to recruit as many as possible centers throughout Germany, to participate in this study. A total sample size of 4000 patients will provide reasonable and valid results for the study aims. The influence of premedication on the primary endpoint change of APAIS-score will be analysed by a multivariable analysis of covariance considering several baseline characteristics. In case of significant interaction terms, subgroup analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Only legally competent patients
* Written informed consent prior to study participation
* Age ≥18 years, both genders
* Elective surgery
* Expected surgery duration ≥ 30 minutes
* Planned general or combined regional and general anaesthesia
* Planned extubation (or removal of airway device) at the end of surgery

Exclusion Criteria:

* Age <18 years
* Non-fluency in German language
* Alcohol and/ or drug abuse
* Chronic benzodiazepine treatment
* Intracranial surgery
* Local or solely regional anaesthesia
* Monitored anaesthesia care/ Sedation
* Cardiac surgery
* Ambulatory surgery
* Repeated surgery with previous participation in the trial
* Expected continuous mandatory ventilation after surgery
* Patients with severe neurological or psychiatric disorders
* Refusal of study participation by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, meeting all inclusion and none exclusion criteria, will be enrolled in the study, independent whether they will receive a premedication or not. The study will be conducted in at least 25-30 German sites.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of the preoperative anxiety level | Up to 30 days
  Change of the preoperative anxiety level, measured with the anxiety measuring scale, named: "Amsterdam Preoperative Anxiety and Information Scale (APAIS)". The measure of agreement with six statements is graded on a 5-point Likert scale from 1 "not at all" to 5 "extremely." A score of ≥11 identify anxious patients in clinical practice. Assessed at: pre-interventional at baseline visit (visit 0) and pre-interventional before surgery (visit 1).

SECONDARY OUTCOMES:
Change in systolic blood pressure | Up to 31 day
  Difference in the haemodynamic variable systolic blood pressure (measured in mmHg) between the assessment pre-interventional at baseline visit (visit 0) and the pre-interventional visit right before surgery (visit 1) and directly post-interventional in the recovery room at visit 2.
Change in diastolic blood pressure | Up to 31 day
  Difference in the haemodynamic variable diastolic blood pressure (measured in mmHg) between the assessment pre-interventional at baseline visit (visit 0) and the pre-interventional visit right before surgery (visit 1) and directly post-interventional in the recovery room at visit 2.
Change in heart rate | Up to 31 day
  Difference in haemodynamic variable (heart rate) between patients with and without premedication. The assessment is conducted pre-interventional at baseline visit (visit 0), in the pre-interventional visit right before surgery (visit 1) and directly post-interventional in the recovery room at visit 2. The values are presented as beats per minute.
Change in oxygen saturation | Up to 31 day
  Difference in the respiratory variable (oxygen saturation) between patients with and without premedication. The assessment is conducted pre-interventional at baseline visit (visit 0), in the pre-interventional visit right before surgery (visit 1) and directly post-interventional in the recovery room at visit 2. The values are presented in percent.
Difference in the cognitive function at baseline as part of the baseline frailty assessment | 1 day
  Cognitive function will be assessed at baseline as part of the frailty assessment according to Oresanya, among the patients who received a premedication and patients without premedication. It will be assessed by the Mini-Cog test, which is a 3-minute instrument that can increase detection of cognitive impairment. It consists of two components, a 3-item recall test for memory and a simply scored clock drawing test.
  Scale: word recall: 0-3 points; Clock Draw: 0 or 2 points; Total Score: 0-5 points
Difference in the medical history at baseline as part of the baseline frailty assessment | 1 day
  Medical history will be assessed at baseline and used for the combined frailty assessment according to Oresanya. Patients will be scored as frail, if ≥ 3 comorbidities are present of the Charlson Comorbidity Index.
Difference in the laboratory value albumin at baseline as part of the baseline frailty assessment | 1 day
  Laboratory value Albumin (unit: g/dl or g/l, depending on the hospital routine), will be assessed according to the clinical routine of the centres. This assessment is optional. It will occur at baseline and will be used for the combined frailty assessment according to Oresanya.
Difference in the laboratory value creatinine at baseline as part of the baseline frailty assessment | 1 day
  Laboratory value Creatinine (unit:mg/dl or µmol/l, depending on the hospital routine), will be assessed according to the clinical routine of the centres. This assessment is optional. It will occur at baseline and will be used for the combined frailty assessment according to Oresanya.
Difference in the laboratory value haemoglobin at baseline as part of the baseline frailty assessment | 1 day
  Laboratory value Creatinine (unit: g/dl or mmol/l, depending on the hospital routine), will be assessed according to the clinical routine of the centres. This assessment is optional. It will occur at baseline and will be used for the combined frailty assessment according to Oresanya.
Difference in the laboratory value haematocrit at baseline as part of the baseline frailty assessment | 1 day
  Laboratory value haematocrit (unit: l/l or %, depending on the hospital routine), will be assessed according to the clinical routine of the centres. This assessment is optional. It will occur at baseline and will be used for the combined frailty assessment according to Oresanya.
Difference in history of falls at baseline as part of baseline frailty assessment | 1 day
  History of falls in the previous 6 months will be assessed at baseline as part of the combined frailty assessment according to Oresanya, among the patients who received a premedication and patients without premedication. Patients will be asked, whether the had one fall, more than one fall, or no fall in the previous 6 months. Patients with more than 1 fall in the last 6 months, has to be marked as "frailty" criterion present according to Oresanya.
Difference in the mobility of the patients as part of baseline frailty assessment | 1 day
  The timed "Up & Go" test, will be used to assess the mobility of the patients at baseline, as part of the frailty assessment according to Oresanya, among the patients who received a premedication and patients without premedication. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Unintentional weight loss at baseline as part of baseline frailty assessment | 1 day
  Unintentional weight loss will be assessed at baseline as part of the frailty assessment. Patients will be asked if they have lost >4,5kg weight in the last year.
Patient satisfaction: Bauer Satisfaction Questionnaire | From intervention up to the 1st postoperative day (visit 3).
  Difference in patients satisfaction about the surgery between patients who received a premedication and patients without premedication, measured with the Bauer Satisfaction Questionnaire (Reference 1) on the first postoperative day (visit 3). Patients rate their satisfaction regarding the first ten questions on a 3 point likert scale, regarding the questions #11 to 15 on a 4 point likert scale and the last question #16 is a yes/no question.
Cognitive recovery | Pre-interventional at baseline visit (visit 0) up to the 1st postoperative day (visit 3).
  Difference in cognitive recovery (defined as difference between baseline assessment and assessment on the first postoperative day) between the two study-groups, measured by the Mini-cog .
Early postoperative delirium | Pre-interventional at baseline visit (visit 0) up to the 1st postoperative day (visit 3).
  Difference in the number of people with a new diagnosed early postoperative delirium between the two study groups, measured with the Confusion Assessment Method (CAM). There will be two assessments (visit 0 and 3).
Perioperative change of sleeping quality: Numeric Rating Scale | Pre-interventional at baseline visit (visit 0) up to the 1st postoperative day (visit 3).
  Difference in the change of the perioperative sleeping quality between the two different study groups, measured with the Numeric Rating Scale (numbers from 0-10) at baseline (visit 0), surgery day pre-operative (visit 1) and first postoperative day (visit 3).
Perioperative change of pain: Numeric Rating Scale | Pre-interventional at baseline visit (visit 0) up to the 1st postoperative day (visit 3).
  Difference in the change of pain between the two different study groups, measured with the Numeric Rating Scale (numbers from 0-10) at baseline (visit 0), surgery day pre-operative (visit 1), surgery day post-operative (visit 2) and first postoperative day (visit 3).
Perioperative change of well-being | Pre-interventional at baseline visit (visit 0) up to the 1st postoperative day (visit 3).
  Difference in the change of the perioperative well-being between the different two study groups, measured with the Numeric Rating Scale (numbers from 0-10) at baseline (visit 0) and first postoperative day (visit 3).
Patient cooperation directly preoperatively | On the day on surgery (1 day)
  Difference in the patient cooperation directly preoperative between the two different study groups, measured with the Numeric Rating Scale (numbers from 0-10).
Patients with rescue-midazolam application before anaesthesia induction | On the day on surgery (1 day)
  Difference in the number of patients who require "rescue-midazolam" application (additional midazolam) before anaesthesia induction between the two study groups.
Time to extubation | At the end of surgery after cessation of the hypnotic agent until extubation (1 day)
  Difference in the needed time to extubation between the two study groups, measured after cessation of the hypnotic agent till removal of endotracheal tube or laryngeal mask airway.
Change in the health-related quality of life assessment: European Quality of Life 5 Dimensions 3 Level questionnaire (EQ-5D-5L) | Pre-interventional at baseline visit (visit 0) up to the 30th day (visit 4) after intervention
  Difference in the change of the health-related quality of life between the two study-groups, measured with the European Quality of Life 5 Dimensions 3 Level questionnaire (EQ-5D-5L). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. For analysis, please refer to the website of the test (please see reference 2)
Longer-term combined outcome of mortality or the new-onset of serious cardiac or pulmonary complications, or acute stroke, or acute kidney | 30 days after intervention (visit 4)
  Difference in the rate of mortality or the new-onset of serious cardiac or pulmonary complications, or acute stroke, or acute kidney injury between the two different study groups, assessed by interview and review of the medical history.
Predefined complications | Surgery day (1 day)
  Difference in the number of predefined complications on the surgery day according to the medical charts between the two different study groups.
Hospital length of stay (LOS) | 30 days after intervention (visit 4)
  Difference in the hospital length of stay (LOS) between the two different study groups.
Intensive care unit length of stay (ICU)-LOS | 30 days after intervention (visit 4)
  Difference in the intensive care unit (ICU)-LOS between the two different study groups.
Patient's functional status of independency | From the baseline visit (visit 0) to the 30th postoperative day (visit 4).
  Difference in the functional recovery between the two study groups, assessed by interview of the patient according to the National Surgical Quality Improvement Program (NSQIP). The questions contain the classification into independent, partially dependent, and totally dependent.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kowark née Stevanovic, MD, Principal Investigator — Department of Anesthesiology, University Hospital Aachen, Germany
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bauer M, Bohrer H, Aichele G, Bach A, Martin E. Measuring patient satisfaction with anaesthesia: perioperative questionnaire versus standardised face-to-face interview. Acta Anaesthesiol Scand. 2001 Jan;45(1):65-72. doi: 10.1034/j.1399-6576.2001.450111.x. PMID 11152036
- [Background] https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-3L_UserGuide_2015.pdf